CLINICAL TRIAL: NCT05884307
Title: Trans Care: An Online Intervention to Reduce Symptoms of Gender Dysphoria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0644: FAA; UW Baldwin Endowment (Other: UW Madison); Protocol Version 11/7/2023 (Other: UW Madison); A171600 (Other: UW Madison)
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gender Dysphoria
Keywords: coping; trans and nonbinary; online intervention; gender minority stress
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans and Nonbinary Adults (Experimental)
  Interventions: Other: Trans Care Web App

INTERVENTIONS:
Other: Trans Care Web App — an educational and interactive website designed to improve coping strategies of TNB individuals

SUMMARY:
The current project aims to improve the well-being of trans and nonbinary (TNB) individuals through an online intervention (Trans Care) targeting the reduction of symptoms of gender dysphoria. The Trans Care intervention will involve the creation of an online intervention comprised of eight modules intended to reduce symptoms of gender dysphoria, increase active coping, and improve the well-being of TNB individuals. Aim 1 is a feasibility and acceptability study of the proposed intervention and will enroll 100 TNB participants to provide feedback to inform a follow-up randomized controlled trial.

DETAILED DESCRIPTION:
The overall purpose of this project is to create a free intervention that can be disseminated widely throughout TNB communities to improve well-being in an easy, accessible way. Development and execution of the Trans Care intervention involves two primary aims:

* Aim 1) Feasibility and acceptability analysis (FAA) [represented by this study record]
* Aim 2) A pilot randomized controlled trial (RCT) of Trans Care's efficacy [to be registered to a separate study record]

Aim 1 involves qualitative and quantitative feedback regarding the content of the Trans Care intervention modules, impact on TNB participants well-being, and feasibility and acceptability of Trans Care intervention. Results from the FAA study will then be analyzed and presented to our community partners who will help us develop modifications to Trans Care to increase its efficacy and ease of use.

Aim 1 Hypotheses:

* The investigators expect that qualitative responses from participants in the FAA study overall will reflect that the Trans Care intervention was feasible and helpful. Any proposed changes from participants' qualitative responses will be incorporated into the final Trans Care intervention presented in the RCT.
* The investigators expect that participants in the FAA study will endorse high scores three scale assessment of feasibility and acceptability.

Aim 1 Endpoints:

The primary endpoint of the study is to determine if the Trans Care intervention is feasible and helpful to TNB individuals for improving their coping strategies. This will be determined through qualitative prompts and a quantitative measure of feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Identify as transgender, transsexual, nonbinary, and/or have a transgender history.
* Experience gender dysphoria.
* Time available to commit to completing a 4-5-hour online intervention and 1-2 hours to complete follow up surveys

Exclusion Criteria:

* under 18 years old
* individual does not identify as transgender, transsexual, nonbinary, and/or have a transgender history
* does not experience gender dysphoria
* is unable to commit to the time requirements of the study
* does not have access to an internet compatible device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) Score | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  The AIM is a 4-item measure of intervention acceptability, each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. Total mean scores range from 1 - 5, higher scores indicate higher acceptability.
Intervention Appropriateness Measure (IAM) Score | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  IAM is a 4-item measure of intervention appropriateness, each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable. A total mean score ranges from 1 - 5, higher scores indicate higher appropriateness.
Feasibility of Intervention Measure (FIM) Score | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  FIM is a 4-item measure of intervention feasibility, each item is rated on a 1-5 scale, with 1 = not at all acceptable and 5 = very acceptable, with a total mean score ranging from 1 to 5, higher scores indicate higher feasibility.
Summary of Qualitative Prompts | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  Participants will be given four prompts to qualitatively assess their experience with the intervention. What you liked most? What would you change? What was most helpful? and What was least helpful?
  Thematic analysis will be conducted to analyze participants' responses to determine predominant changes suggested by participants
Trans Care Intervention Specific Feasibility and Acceptability Score | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  This measure is score from 0 to 4 in each of 5 domains: overall assessment, helpfulness, instructions, videos, and activities. Higher scores indicate higher feasibility and acceptability.
Digital Working Alliance Inventory (D-WAI) Score | post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  The D-WAI is scored from 7-point Likert-type scale from 1 (strongly disagree) to 7 (strongly agree), for a total range of scores from 7-42 where higher scores indicate higher perceived app effectiveness.

SECONDARY OUTCOMES:
Depression, Anxiety, and Stress Scale (DASS-21) Score | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  DASS-21 is scored from 0-3 in each of 3 domains: depression, anxiety, and stress. Higher scores mean increased depression, anxiety, and stress.
Gender Congruence and Life Satisfaction Scale (GCLS) Score | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  GCLS asks participants to think about how they have felt over the last 6 months. Responses are scored on a 5-point Likert scale (always = 1; never = 5). A higher scores mean greater gender congruence, greater gender-related well-being, and greater life satisfaction.
Modified Gender Minority Stress and Resilience Measure (M-GMSRM) Score | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  M-GMSRM is scored from 0-100 where higher scores indicate higher stress.
Trans and Nonbinary Coping Measure (TNCM) Score | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  TNCM is scored from 0-5 where higher scores indicate greater frequency of utilization of coping strategy in each of 6 domains: Social Support / Connection, Social Activism, Hope, Strategic Gender Expression, Behavioral Avoidance, Identity Non-Disclosure.
Brief Cope Score | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  The Brief Cope survey is scored from 1-4 in each of 3 domains: problem-focused coping, emotion-focused coping, and avoidant-coping. Higher scores indicate increased coping mechanisms.
Alcohol Use Disorder Identification Test | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  This is scored from 0-40 where higher scores are indicative of increased dependence on alcohol.
Number of Days in the Past Week You Consumed Alcohol | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  7 = 7 days, 6 = 6 days, 5 = 5 days, 4 = 4 days, 3 = 3 days, 2 = 2 days, 1 = 1 day, 0 = no days
Quantity of Alcohol Use | baseline and post intervention (intervention can take up to 5 hours to complete, participant has up to 1 month to complete it)
  How many alcoholic drinks, on average, have you had per day during the past week? An alcoholic drink is defined as 1 beer, 1 glass of wine, 1 shot of alcohol, or 1 mixed drink.
  Response options:
  5 = 12+ drinks, 4 = 8-11 drinks, 3 = 5-7 drinks, 2 = 3-4 drinks, 1 = 1-2 drinks, 0 = none

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Budge, PhD, LP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Hypothesis and Design Plan Pre-registered on OSF — https://osf.io/ebq6w